CLINICAL TRIAL: NCT04703881
Title: Tolerance and Acceptability Evaluation AYMES ActaGain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aymes International Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AY-ActaGain
Record Dates: First submitted 2021-01-05; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AYMES ActaGain (Experimental): Patients of the intended target group (e.g. MUST score ≥ 1, with or at risk of disease related malnutrition) with an anticipated period of nutritional support ≥ 4 weeks will be changed / started on an equivalent prescription of 'AYMES ActaGain' for a period of 30 days.
  Interventions: Dietary Supplement: AYMES ActaGain

INTERVENTIONS:
Dietary Supplement: AYMES ActaGain — AYMES ActaGain is a Food for Special Medical Purposes (FSMP) and must, therefore, be used under medical supervision. It is designed as a supplement to the diet but can also be used as a sole source of nutrition.

SUMMARY:
To evaluate tolerance and acceptability of 'AYMES ActaGain' in patients requiring supplementary oral nutritional support compared with currently available alternatives.

DETAILED DESCRIPTION:
To evaluate tolerance and acceptability of 'AYMES ActaGain' in patients requiring supplementary oral nutritional support compared with currently available alternatives, measuring outcomes of GI effects, Compliance, product preference, convenience etc.

To obtain data to support an ACBS submissions for 'AYMES ActaGain' (to allow for prescription in the community at NHS expense).

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients.
* ≥ 18 years of age.
* Patients of the intended target group (e.g. MUST score ≥ 1, with or at risk of disease related malnutrition) with an anticipated period of nutritional support ≥ 4 weeks.
* Patient is able and willing to provide written informed consent.

Exclusion Criteria:

* Patients with medical or dietary contraindication to any feed ingredients.
* Patients requiring sole enteral tube feeding or parenteral nutrition.
* Patients with chronic renal disease requiring dialysis.
* Patients with liver failure.
* Patients for whom the investigator has concerns regarding the ability or willingness of the patient and or carer to comply with protocol requirements.
* Patients assessed by a Speech and Language Therapist who require thickened fluids.
* Participation in any other studies that may interfere with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Gastro-Intestinal Tolerance when consuming AYMES ActaGain | 30 days
  To assess gastro-intestinal tolerance of 'AYMES ActaGain' in patients in the community requiring oral nutritional supplementation. Monitoring includes recording the number of any GI complaints via a daily diary.

SECONDARY OUTCOMES:
Acceptability and Palatability of Consuming the Nutritional Supplement: questionnaire | 30 days
  To assess the acceptability of 'AYMES ActaGain' in patients in the community requiring oral nutritional supplementation. At the end of the intervention period an acceptability and preference questionnaire will be completed by the patient in order to seek their opinion on the taste, smell, texture and overall liking of the new supplement drink. A 5 point hedonic scale will be used.
Compliance | 30 days
  To assess the acceptability of 'AYMES ActaGain' in patients in the community requiring oral nutritional supplementation. A daily compliance diary will be kept detailing compliance to prescription versus prescribed amount.

CONTACTS AND LOCATIONS:
Locations (1):
- AYMES International Ltd., Haywards Heath, United Kingdom

IPD SHARING:
Plan to Share IPD: No